CLINICAL TRIAL: NCT01344135
Title: Cost Effectiveness Analysis and Clinical Outcome of Nutritional Rehabilitation on Physical Functioning and Cardiometabolic Risk Profile in COPD Patients With Muscle Atrophy
Brief Title: Nutritional Rehabilitation in Chronic Obstructive Pulmonary Disease (COPD) Patients With Muscle Atrophy
Acronym: NUTRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: The Netherlands Asthma Foundation (Other); Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MEC 11-3-004
Record Dates: First submitted 2011-04-12; First posted 2011-04-28 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2011-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Muscular Atrophy
Keywords: Pulmonary Disease, Chronic Obstructive; Muscular Atrophy; Nutritional rehabilitation; Counselling
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Muscular Atrophy | interventions — Dietary Supplements; Counseling; Motivational Interviewing; Exercise; Accelerometry

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (placebo control) (Placebo Comparator): 60 clinically stable COPD patients with muscle atrophy, eligible for out-patient pulmonary rehabilitation
  Interventions: Dietary Supplement: Placebo supplement; Behavioral: Feedback on physical activity level
- Group 2 (nutritional intervention) (Experimental): 60 clinically stable COPD patients with muscle atrophy, eligible for out-patient pulmonary rehabilitation
  Interventions: Dietary Supplement: Dietary supplementation; Behavioral: Nutritional counselling; Behavioral: Feedback on physical activity level

INTERVENTIONS:
Dietary Supplement: Dietary supplementation — Phase A, Rehabilitation (4 months): 3 nutritional supplements daily
  Phase B, Maintenance (8 months): nutritional supplementation on advice (1 supplement daily)
  Phase C, Follow-up (3 months): no supplementation
  Other Names: Nutritional supplementation; Dietary supplement; Nutritional supplement; Food supplement
  Arms: Group 2 (nutritional intervention)
Dietary Supplement: Placebo supplement — Phase A, Rehabilitation (4 months): 3 placebo nutritional supplements daily
  Phase B, Maintenance (8 months): No supplementation
  Phase C, Follow-up (3 months): No supplementation
  Other Names: Non-active supplement
  Arms: Group 1 (placebo control)
Behavioral: Nutritional counselling — Phase A, Rehabilitation (4 months): No counselling
  Phase B, Maintenance (8 months): Nutritional counselling (4x)
  Phase C, Follow-up (3 months): No counselling
  Aim:
  1. Optimising dietary intake to physical activity pattern and energy expenditure.
  2. Minimize deterioration of dietary intake during acute exacerbations.
  3. Optimize dietary lipid profile with respect to total fat intake; trans fatty acids and proportion of poly-unsaturated fatty acids to modulate cardiovascular risk and muscle fatty acid metabolism.
  4. Increasing adherence/compliance by addressing issues like taste fatigue, gastro-intestinal symptoms, individual preferences and lifestyle.
  Other Names: Counselling; Motivational interviewing; Increasing self-regulation skills; Increasing perceived competence and autonomy
  Arms: Group 2 (nutritional intervention)
Behavioral: Feedback on physical activity level — Phase A, Rehabilitation (4 months): No exercise counselling
  Phase B, Maintenance (8 months): Exercise counselling (2x)
  Phase C, Follow-up (3 months): No exercise counselling
  Aim:
  1. Integration of exercise behaviour into daily routine
  2. Improvement of self-regulation skills (e.g. self-monitoring, goal setting, action planning)
  3. Increasing adherence/compliance by addressing issues like coping with difficult situation, individual preferences and lifestyle
  Other Names: Exercise; Accelerometry

SUMMARY:
To study in clinically stable Chronic Obstructive Pulmonary Disease (COPD) patients with muscle atrophy:

1. The short-term effects of 4 months exercise training including nutritional supplementation versus exercise training alone on physical functioning (skeletal muscle strength and exercise capacity) and body composition.
2. The long-term effects of 4 months of exercise training and nutritional supplementation followed by 8 months of nutritional counseling (with supplementation on advice) and feedback on physical activity level versus 4 months of exercise training and 8 months with feedback on physical activity level alone on physical functioning, body composition and cardiometabolic risk profile;
3. The cost-effectiveness of exercise rehabilitation and nutritional intervention versus exercise rehabilitation alone.

DETAILED DESCRIPTION:
Rationale. Recent guidelines state that pulmonary rehabilitation should be part of integrated care of patients with COPD and not limited to end stage disease. The investigators hypothesize that clinically stable COPD patients muscle atrophy, irrespective of the severity of airflow obstruction, show more pronounced long-term improvement in physical functioning and cardiometabolic risk profile after a rehabilitation programme including nutritional intervention (supplementation and counseling) than after a pulmonary rehabilitation programme without nutritional intervention, at acceptable costs. Nutritional supplementation focuses on enhancing the efficacy of the exercise training. Nutritional counseling aims at maintaining energy balance and modulating cardiovascular disease risk.

Study design. The research aims will be addressed in a multi-centre, randomized, clinical trial.

Phase A, Rehabilitation (4 months):

* Group 1: Supervised exercise training and 3 placebo nutritional supplements daily
* Group 2: Supervised exercise training and 3 nutritional supplements daily

Phase B, Maintenance (8 months):

* Group 1: Exercise counseling (2x)
* Group 2: Exercise counseling (2x), nutritional counseling (5x) (and 1 nutritional supplement a day on indication)

Phase C, Follow-up (3 months):

* Group 1: no intervention
* Group 2: 1 nutritional supplement a day on request

Nature and extent of the burden and risks associated with participation and benefits. This study aims to tailor pulmonary rehabilitation. Participants of group 1 are visiting their rehabilitation centre 3 times for study related measurements within 15 months (2 times feedback on physical activity, 1 measurement visit). Participants of group 2 will be asked to visit their rehabilitation centre for 6 times (1 measurement visit, 3 times nutritional counseling, 1 time for feedback on physical activity, 1 time for nutritional counseling and feedback on physical activity combined) within 15 months. For both groups baseline measurements and outcome measurements after rehabilitation are already included in the CIRO rehabilitation programme.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Obstructive Pulmonary Disease
* Muscle atrophy (a FFMI under the sex- and age-specific 25th percentile FFMI values, assessed by DEXA)
* Eligible for pulmonary rehabilitation

Exclusion Criteria:

* COPD patients under the age of 18;
* Allergy or intolerance to fish, milk or other components of the study product;
* Investigator's uncertainty about the willingness or ability of the patient to comply with the protocol requirements;
* Not able to stop current supplement use or if total use will be above safe upper limits;
* Participation in any other study involving investigational or marketed products concomitantly or within two weeks prior to entry into the study;
* Pregnancy;
* Life threatening diseases like tuberculosis, carcinoma, AIDS (including HIV+), acute leukaemia etc.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle strength | 0, 12 months
  Skeletal muscle strength assessed by isokinetic dynamometry (Biodex®)

SECONDARY OUTCOMES:
Cardiometabolic risk profile | 0, 4, 12 months
  * lipid profile (blood)
  * systemic inflammatory profile (blood)
  * blood pressure(hematometer)
  * HOMA index (blood)
  * visceral fat mass (DEXA)
  * AGEs skin (AGE reader)
Health related quality of life | 0, 4, 12, 15 months
  Assessed by:
  * SGRQ: Saint George Respiratory Questionnaire
  * SF36: Short Form - 36
  * EQ5D: EuroQol 5 domains, extended with energy/fatique domain
Dyspnoea | 0, 4, 12, 15 months
  Assessed by:
  -MRC-index: Medical Research Council dyspnoea scale
Body composition | 0, 4, 12 months
  Assessed by
  - DEXA scan
Exercise capacity | 0, 4, 12 months
  Assessed by:
  - Constant Work Rate Test (CWRT)
Plasma levels of supplemented (micro)nutrients | 0, 4, 12 months
  Assessed by:
  * Plasma amino acids (leucine)
  * Vitamin D (plasma calcidiol 25(OH)D )
Bone mass density | 0, 4, 12 months
  Assessed by:
  - DEXA scan
Physical activity | 0, 4, 12, 15 months
  Assessed by:
  - Accelerometry

CONTACTS AND LOCATIONS:
Overall Officials: Annemie Schols, Prof., Study Director — Maastricht UMC+ / NUTRIM, Respiratory Medicine; Maureen Rutten, Dr., Principal Investigator — Erasmus Medical Centre, Institute for Medical Technology Assessment; Emiel FM Wouters, Prof., Principal Investigator — Maastricht UMC+ and CIRO, Respiratory Medicine
Locations (1):
- CIRO, Horn, Limburg, Netherlands